CLINICAL TRIAL: NCT01075581
Title: Hemostatic and Hemodynamic Effects of Intranasal Injection Compared to Topical Administration of Epinephrin in Endoscopic Sinus Surgery
Brief Title: Intranasal Injection Versus Topical Administration of Epinephrin During Endoscopic Sinus Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr Roee Landsberg, The Ear, Nose and Throat (ENT) Department - Head and Neck Surgery at the Tel Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-10-RL-0035-CTIL
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Hypertension; Hypotension; Tachycardia; Bradycardia; Arrhythmia
Keywords: Hemodynamic instability; Hemostasis
MeSH Terms: conditions — Hypertension; Hypotension; Tachycardia; Bradycardia; Arrhythmias, Cardiac | interventions — Epinephrine; Administration, Topical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical administration (Active Comparator): An an intranasal injection of saline will be used as control, and thereafter cotton pledgets soaked in 1 mL epinephrine 1:1,000 will be placed in the nasal cavity during surgery when necessary.
  Interventions: Drug: Epinephrin (Topical administration)
- Intranasal injection (Experimental): An intranasal injection of 8 mL epinephrine 1:100,000 will be performed as traditionally practiced in ESS. Thereafter, cotton pledgets soaked in 1 mL epinephrine 1:1,000 will be placed in the nasal cavity during surgery when necessary.
  Interventions: Drug: Epinephrin (Intranasal injection)

INTERVENTIONS:
Drug: Epinephrin (Intranasal injection) — A total of 8 mL of epinephrine 1:100,000 will be injected in the lateral nasal wall, followed by placement of cotton pledgets (soaked in 1 mL epinephrine 1:1,000) in the nasal cavity when required.
  Other Names: Adrenaline
  Arms: Intranasal injection
Drug: Epinephrin (Topical administration) — An intranasal injection of saline solution, followed by placement of cotton pledgets (soaked in 1 mL epinephrine 1:1,000) in the nasal cavity when required.
  Other Names: Adrenaline
  Arms: Topical administration

SUMMARY:
Intranasal injection of epinephrine is used routinely during endoscopic sinus surgery (ESS) to reduce bleeding in the nasal mucosa and thereby improve visualization of the surgical field. However, systemic absorption of epinephrine via the nasal mucosa is often accompanied by cardiovascular side effects during the early postinjection period, putting in risk patients with cardiovascular morbidity. Evidence indicate that topical administration of epinephrine achieves similar hemostatic effects compared with injection of epinephrine, while avoiding systemic adverse effects. We wish to conduct a prospective controlled trial assessing the hemostatic and hemodynamic effects of intranasal injection compared to topical application of epinephrin during ESS, in order to evaluate whether the previous could be avoided due to its untoward effects.

We hypothesize that topical administration of epinephrine provides a hemostatic effect not inferior to that of intranasal injection while minimizing hemodynamic instability during ESS.

DETAILED DESCRIPTION:
Introduction:

Intranasal injection of epinephrine is used routinely during endoscopic sinus surgery (ESS) to reduce bleeding in the nasal mucosa and hence improve visualization of the surgical field [1, 2].

Systemic absorption of epinephrine via the nasal mucosa, due to its vasoconstriction ability and cardiac effect, is often accompanied by cardiovascular side effects (e.g., hypertension, hypotension, tachycardia, cardiac arrhythmias, etc) during the early postinjection period [1, 3-5]. In patients with minimal cardiac reserve, these acute hyperdynamic effects may result in myocardial ischemia or infarction [6, 7]. The nasal mucosa has an excellent absorbing capability which may be utilized for local administration of vasoconstrictive substances instead of intranasal injection [8, 9], thus avoiding their systemic adverse effects .

Evidence indicate that topical use of epinephrine may achieve similar hemostatic effects compared with injection of epinephrine [10]. Another pilot study has demonstrated that epinephrine injection better facilitates visualization of the surgical field, yet topical application does not involve hemodynamic side effects [11]. However, a prospective, randomized larger trial has shown that, when local anesthetic containing epinephrine was used compared with normal saline (NS) injection for ESS, there was no significant reduction in intraoperative blood loss or duration of surgery. More importantly, a significantly higher mean arterial blood pressure (MABP) was associated with injection of epinephrine [2].

The objective of the current study is to compare the hemostatic and hemodynamic effects of intranasal injection versus topical application of epinephrin during ESS, in order to evaluate whether the previous could be avoided due to its untoward effects.

Study design:

After obtaining informed consent, patients will be assigned to one of two groups - intranasal injection group (IG) or topical application (TG) of epinephrine, by computer-generated assignment of random numbers.

Intra-operative surgical management:

Routine ESS will be performed on each subject. Resection and removal of different structures in the sinonasal complex will be executed appropriately as indicated according to underlying pathology.

Intra-operative vasoconstrictor administration Vials containing either epinephrine 1:100,000 or saline will be prepared in the operating room (OR) by the surgeon, with the assistance of the OR nurse. The content of the vials will not be disclosed to the surgeon (or anesthetist), who will thus not be aware of the type of solution being diluted. While patients allocated to the IG group will be injected with epinephrine, saline injection (total of 8 mL) will be used in the TG group.

Topical epinephrine will be applied in exactly the same manner and quantity for the saline-injected group as for the IG group:

Following initiation of general anesthesia and intubation, cotton pledgets soaked in 1 mL epinephrine 1:1,000 will be positioned in the nasal cavity for approximately 10 minutes. Following this, all patients will receive intranasal injection according to their assigned group. In the IG group a total of 8 mL of epinephrine 1:100,000 will be injected in the lateral nasal wall in two locations: the area superior to the insertion of the middle turbinate and area anterior to the posterior insertion of the middle turbinate, at the spheno-palatine artery region. The injection will be applied to both sides (total of 8 mL). Following the injection, Epinephrine-soaked cotton pledgets (1 mL of 1:1,000) will be placed at the middle meatus and anterior to the sphenoethmoidal recess. During the procedure the pledgets will be used at various locations as required for primary decongestion.

In the TG group, saline will be injected instead of epinephrine.

Patient assessment:

Patients' parameters will be collected during the procedure by an anesthesiologist via iMDsoft software. A printout delineating the following data will be obtained: heart rate, ECG for arrhythmias, systolic (SP) and mean arterial pressure (MAP) measured from a blood pressure cuff once per 2 minutes, and total intraoperative blood loss. These parameters will be monitored by the anesthetist throughout the procedure.

Study patients will be monitored throughout the procedure for any hemodynamic events potentially related to the vasoconstrictor applied to them. We will continue follow-up until they discharge in order to detect any post-operative complications that may occur due to systemic absorption of epinephrine.

Previous studies have demonstrated a significant increase in the plasma catecholamine level after nasal injection of epinephrine, which was associated with hemodynamic fluctuations [1, 11]. We therefore wish to analyze the systemic absorption of injected epinephrine during ESS.

Intraoperative catecholamine blood levels (epinephrine and norepinephrine) will be obtained by taking blood samples (7ml in each sample) from each patient: immediately after intubation (baseline), before pladget placement, 5min after pladget placement, before injection (approximately 10 minutes after applying epinephrine gauze strips), 2min post injection and placement of cotton pledgets (to both sides), 5min, 10min and 15 minutes post injection.

Other records will include: patient demographics, the duration of surgery, extent of nasosinusal polyposis/number of structures to be operated, the presence of polyps will be recorded, and need for intraoperative pharmacological intervention (vasopressors, vasodilators, inotropes, etc.).

The primary endpoint of the study will be changes in intraoperative hemodynamic parameters, and incidence of hemodynamic events during surgery, and specifically in the immediate post injection/topical application period (5min). These will include:

1. Lowest and highest HR, SP and MAP values.
2. Mean HR, SP and MAP during surgery.
3. Incidence of hypotensive and hypertensive events (>20% relative to baseline).
4. Incidence of tachycardic (HR>115) and bradycardic (HR<55) events. Analysis for correlation of these parameters with catecholamine blood levels will be performed.

The secondary endpoints will include:

1. Extent of nasal bleeding (estimated by assessment of the suction bottles, sponges, and the surgical drapes and gowns).
2. The total number of epinephrin pledgets used during surgery.
3. Incidence of arrhythmias and ST changes on ECG.
4. Subjective surgeons' evaluation of the feasibility of performing the procedure, effectiveness of hemostasis, and visualization of the operative field.
5. Pharmacokinetics of epinephrine administered to the nasal mucosa via injection and topical administration.
6. Post-operative complications due to systemic absorption of epinephrine in patients with risk factors (i.e., arteriosclerosis, hypertension, ischemic heart disease and other cardiac problems, anemia, preexistent liver or renal damage, and endocrinologic dysfunction such as hyperthyroidism, phaeochromocytoma, and diabetes mellitus) will be monitored until the patients discharge.

References

1. Anderhuber W, Walch C, Nemeth E, Semmelrock HJ, Berghold A, Ranftl G, Stammberger H. Plasma adrenaline concentrations during functional endoscopic sinus surgery. Laryngoscope 1999;109: 204-7.
2. Javer AR, Gheriani H, Mechor B, Flamer D, Genoway K, Yunker WK. Effect of intraoperative injection of 0.25% bupivacaine with 1:200,000 epinephrine on intraoperative blood loss in FESS. Am J Rhinol Allergy 2009;23: 437-41.
3. van Hasselt CA, Low JM, Waldron J, Gibb AG, Oh TE. Plasma catecholamine levels following topical application versus infiltration of adrenaline for nasal surgery. Anaesth Intensive Care 1992;20: 332-6.
4. Yang JJ, Wang QP, Wang TY, Sun J, Wang ZY, Zuo D, Xu JG. Marked hypotension induced by adrenaline contained in local anesthetic. Laryngoscope 2005;115: 348-52.
5. Moshaver A, Lin D, Pinto R, Witterick IJ. The hemostatic and hemodynamic effects of epinephrine during endoscopic sinus surgery: a randomized clinical trial. Arch Otolaryngol Head Neck Surg 2009;135: 1005-9.
6. Campagni MA, Howie MB, White PF, McSweeney TD. Comparative effects of oral clonidine and intravenous esmolol in attenuating the hemodynamic response to epinephrine injection. J Clin Anesth 1999;11: 208-15.
7. Kaufman E, Garfunkel A, Findler M, Elad S, Zusman SP, Malamed SF, Galili D. [Emergencies evolving from local anesthesia]. Refuat Hapeh Vehashinayim 2002;19: 13-8, 98.
8. Lang S, Rothen-Rutishauser B, Perriard JC, Schmidt MC, Merkle HP. Permeation and pathways of human calcitonin (hCT) across excised bovine nasal mucosa. Peptides 1998;19: 599-607.
9. Roth Y, Chapnik JS, Cole P. Feasibility of aerosol vaccination in humans. Ann Otol Rhinol Laryngol 2003;112: 264-70.
10. Lee TJ, Huang CC, Chang PH, Chang CJ, Chen YW. Hemostasis during functional endoscopic sinus surgery: the effect of local infiltration with adrenaline. Otolaryngol Head Neck Surg 2009;140: 209-14.
11. Cohen-Kerem R, Brown S, Villasenor LV, Witterick I. Epinephrine/Lidocaine injection vs. saline during endoscopic sinus surgery. Laryngoscope 2008;118: 1275-81.
12. Dershwitz M, Hoke JF, Rosow CE, Michalowski P, Connors PM, Muir KT, Dienstag JL. Pharmacokinetics and pharmacodynamics of remifentanil in volunteer subjects with severe liver disease. Anesthesiology 1996;84: 812-20.
13. Wormald PJ, van Renen G, Perks J, Jones JA, Langton-Hewer CD. The effect of the total intravenous anesthesia compared with inhalational anesthesia on the surgical field during endoscopic sinus surgery. Am J Rhinol 2005;19: 514-20.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA I-III,
* Patients undergoing elective FESS at Sourasky Medical Center for Chronic rhinosinusitis with or without polyposis, including FESS combined with septoplasty and/or conchotomy.

Exclusion Criteria:

* Patients scheduled for endoscopic resection of a tumor or closure of a cerebrospinal fluid leak, and
* Patients for whom epinephrine was contraindicated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hemodynamic alterations (instability) | duration of surgery
  Changes in intraoperative hemodynamic parameters will be monitored continuously,and any event will be documented, including: lowest and highest HR, SP and MAP values; mean HR, SP and MAP during surgery; incidence of hypotensive and hypertensive events (>20% relative to baseline); incidence of tachycardic (HR>115) and bradycardic (HR<55) events.

SECONDARY OUTCOMES:
Hemostasis | duration of surgery
  Hemostatic effects will be evaluated by the following parameters:
  1. By the surgeon, via a subjective surgical grade scoring system.
  2. By the extent of nasal bleeding (estimated by assessment of the suction bottles, sponges, and the surgical drapes and gowns).
  3. By the total number of epinephrin pledgets used during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Roee Landsberg, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel